CLINICAL TRIAL: NCT05144399
Title: Accelerated Treatment of Endocarditis
Acronym: POET II
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Kasper Iversen, Associate professor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18028566
Record Dates: First submitted 2019-08-16; First posted 2021-12-03 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated antibiotic treatment (Experimental): Patients are treated shorter than usual
  Interventions: Other: Accelerated antibiotic treatment
- Standard length of antibiotic treatment (Other): Patients are receiving the standard length of antibiotic treatment
  Interventions: Other: Standard treatment length

INTERVENTIONS:
Other: Accelerated antibiotic treatment — E. faecalis uncomplicated: 4 weeks.
  E. faecalis complicated: 4 weeks.
  S. aureus uncomplicated: 2 weeks.
  S. aureus complicated: 4 weeks.
  Streptococci spp. NVE: 2 weeks.
  Streptococci spp. PVE or abscess: 3 weeks.
  Subsequent to cardiac surgery with a negative valve culture (organism NOT grown in laboratory from valve): Minimum 1 week after surgery regardless of previous antibiotic treatment received.
  Subsequent to cardiac surgery with a positive valve culture (organism grown in laboratory from valve): treatment will continue with the start date of antibiotics changed to the date of surgery.
  Complicated IE defined as patients with abscess, embolic event, surgically treated IE, and/or PVE.
  NVE: native valve endocarditis, PVE: prosthetic valve endocarditis.
  Arms: Accelerated antibiotic treatment
Other: Standard treatment length — E. faecalis uncomplicated: 6 weeks.
  E. faecalis complicated: 6 weeks.
  S. aureus uncomplicated: 4 weeks.
  S. aureus complicated: 6 weeks.
  Streptococci spp. NVE: 4 weeks.
  Streptococci spp. PVE or abscess: 6 weeks.
  Subsequent to cardiac surgery with a negative valve culture (organism NOT grown in laboratory from valve): Minimum 2 weeks after surgery regardless of previous antibiotic treatment received.
  Subsequent to cardiac surgery with a positive valve culture (organism grown in laboratory from valve): treatment will continue with the start date of antibiotics changed to the date of surgery.
  Complicated IE defined as patients with abscess, embolic event, surgically treated IE, and/or PVE.
  NVE: native valve endocarditis, PVE: prosthetic valve endocarditis.
  Arms: Standard length of antibiotic treatment

SUMMARY:
Existing guidelines recommend a duration of antibiotic treatment of endocarditis of 4-6 weeks one or more types of intravenously administered antibiotics. The long hospitalization increases several risks for the patient, including mental strain and increased loss of function. Furthermore, it poses a significant financial burden on the health systems. Current guidelines fail to use available clinical and paraclinical, data collected from patients (echo, temperature, CRP, leukocytes, procalcitonin etc.) to determine duration of treatment. A strategy including these data in treatment algorithms ensures an individualized treatment, targeting the individual patient's course and response to treatment. Thus, the purpose of this open-label, prospective, non-inferiority, RCT study is to investigate the safety and effectiveness of shortening treatment of endocarditis based on the individual patient's initial treatment response, sampling 475 patients, approx. 125 patients with each type of bacteria (Streptococci; Enterococcus faecalis; Staphylococcus aureus).

ELIGIBILITY:
Inclusion Criteria:

* Admitted with left-sided infectious endocarditis (duke criteria)
* < 14 days of relevant antibiotic treatment for endocarditis
* One of the following bacteria: Streptococci, enterococcus faecalis, staphylococcus aureus
* > 18 years old

Exclusion Criteria:

* Known immune incompetency,
* Relapse endocarditis with 6 months,
* Unable to give informed concent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Combined safety endpoint of: All cause mortality, embolic episodes, not planned Heart surgery | 6 months after randomization
  The primary endpoint is a combined endpoint consisting of the following events occurring within six months after the earliest time of potential treatment discontinuation: Death; Embolisms; Heart surgery not planned at the time of randomization.
Primary efficacy endpoint: Difference in number of days alive without antibiotic treatment for endocarditits and/or bacteremia between the two study groups | 6 months after randomization
  The primary efficacy endpoint is the difference in number of days alive without antibiotic treatment for endocarditits and/or bacteremia between the two study groups, assessed from and until 6 months after randomization.

SECONDARY OUTCOMES:
Expenses associated with admission and treatment | 6 months after randomization
  Combined endpoint consisting of expenses due to i admission ii medication iii transportation iv surgery v imaging vi home care
Duration of admission | 6 months after randomization
  Duration of admission
Duration of antibiotic treatment | 6 months after randomization
  Duration of antibiotic treatment
Frequency of catheter complication | 6 months after randomization
  Frequency of catheter complication
Unplanned Heart surgery | 6 months after randomization
  • Unplanned cardiac valve surgery defined as any cardiac surgery which is not planned at the time of randomization. Data will be extracted from the electronic patient journal.
All cause mortality | 6 months after randomization
  All cause mortality
Embolic events | 6 months after randomization
  Embolic events
Re-bacteremia with the primary pathogen | 6 months after randomization
  • Relapse of bacteremia defined as a positive blood culture with the same microorganism as during the initial IE admission (streptococci spp., S. aureus, or E. faecalis). Data will be extracted from the electronic patient journal.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshositalet, Copenhagen
  - Herlev Hospital, Herlev

IPD SHARING:
Plan to Share IPD: No